CLINICAL TRIAL: NCT05424614
Title: Capital's Funds for Health Improvement and Research
Brief Title: Study on the Prognostic Prediction Model of Patients With Acute Intracerebral Hemorrhage by Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-2-1074
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Hemorrhage; Prognosis; Artificial Intelligence
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intracerebral hemorrhage group: Patients with the intracerebral hemorrhage who presented to the hospital within 24 hours of symptom onset
  Interventions: Other: Functional outcome follow-up of patients

INTERVENTIONS:
Other: Functional outcome follow-up of patients — Patients were followed up by telephone after discharge, every 4 weeks, until the end of the 3-month follow-up. Their functional status was determined based on the MRS score (modified Rankin Scale). Those with less than 3 points were defined as having a good prognosis, and those with more than 3 points were defined as having a poor prognosis

SUMMARY:
Spontaneous intracerebral hemorrhage(SICH) is the most lethal and disabling stroke. Timely and accurate assessment of patient prognosis could facilitate clinical decision making and stratified management of patients and is important for improving patient clinical prognosis. However, current studies on the prediction of prognosis of patients with SICH are limited and only include a single variable, with less precise results and inconvenient clinical application, which may lead to delays in effective patient treatment. Our group's previous studies on SICH showed that hematoma heterogeneity and the degree of contrast extravasation within the hematoma are closely related to the clinical outcome of patients, but they are difficult to describe quantitatively based on imaging signs. Based on this, we propose to use radiomics to quantitatively extract hematoma features from NCCT and CTA images, combine them with patients' clinical information and laboratory tests, study their relationship with the prognosis of cerebral hemorrhage, and use artificial intelligence to establish a rapid and accurate prognostic prediction model for patients with SICH, which is of great significance to guide clinical individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. aged 18-80 years; 2. patients diagnosed with acute cerebral hemorrhage by CT examination; 3. complete non-contrast CT and CTA images; 4. the time interval from onset to the first baseline CT and CTA examination is less than 6 hours; 5. follow-up data within 3 months; 6. agree and sign a written document.

Exclusion Criteria:

* 1. Patients with secondary aneurysm hemorrhage; 2. Patients with secondary hemorrhage of cerebrovascular malformation; 3. Patients with dissecting aneurysm hemorrhage; 4. Patients with cerebral infarction hemorrhage transformation; 5. Patients lost to follow-up within 3 months; 6. CT or CTA images have a heavy artefact.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute cerebral hemorrhage (within 6 hours of the onset of symptoms) who presented to the hospital between May 2022 and September 2024 and had complete medical records.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
patient outcome | 3 month
  Neurological recovery status was measured by the modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Shengjun Sun, Principal Investigator — Beijing Neurosurgical Instuitute
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
To obtain individual participant data, please contact the principal investigator.

REFERENCES:
- [Background] Pszczolkowski S, Manzano-Patron JP, Law ZK, Krishnan K, Ali A, Bath PM, Sprigg N, Dineen RA. Quantitative CT radiomics-based models for prediction of haematoma expansion and poor functional outcome in primary intracerebral haemorrhage. Eur Radiol. 2021 Oct;31(10):7945-7959. doi: 10.1007/s00330-021-07826-9. Epub 2021 Apr 16. PMID 33860831
- [Background] Xie H, Ma S, Wang X, Zhang X. Noncontrast computer tomography-based radiomics model for predicting intracerebral hemorrhage expansion: preliminary findings and comparison with conventional radiological model. Eur Radiol. 2020 Jan;30(1):87-98. doi: 10.1007/s00330-019-06378-3. Epub 2019 Aug 5. PMID 31385050
- [Background] Guo R, Zhang R, Liu R, Liu Y, Li H, Ma L, He M, You C, Tian R. Machine Learning-Based Approaches for Prediction of Patients' Functional Outcome and Mortality after Spontaneous Intracerebral Hemorrhage. J Pers Med. 2022 Jan 14;12(1):112. doi: 10.3390/jpm12010112. PMID 35055424
- [Background] Gregorio T, Pipa S, Cavaleiro P, Atanasio G, Albuquerque I, Chaves PC, Azevedo L. Prognostic models for intracerebral hemorrhage: systematic review and meta-analysis. BMC Med Res Methodol. 2018 Nov 20;18(1):145. doi: 10.1186/s12874-018-0613-8. PMID 30458727
- [Background] Fu F, Sun S, Liu L, Gu H, Su Y, Li Y. Iodine Sign as a Novel Predictor of Hematoma Expansion and Poor Outcomes in Primary Intracerebral Hemorrhage Patients. Stroke. 2018 Sep;49(9):2074-2080. doi: 10.1161/STROKEAHA.118.022017. PMID 30354984
- [Background] Wang J, Wang W, Liu Y, Zhao X. Associations Between Levels of High-Sensitivity C-Reactive Protein and Outcome After Intracerebral Hemorrhage. Front Neurol. 2020 Oct 6;11:535068. doi: 10.3389/fneur.2020.535068. eCollection 2020. PMID 33123072
- [Background] Menon G, Johnson SE, Hegde A, Rathod S, Nayak R, Nair R. Neutrophil to lymphocyte ratio - A novel prognostic marker following spontaneous intracerebral haemorrhage. Clin Neurol Neurosurg. 2021 Jan;200:106339. doi: 10.1016/j.clineuro.2020.106339. Epub 2020 Oct 28. PMID 33183885
- [Background] Morotti A, Arba F, Boulouis G, Charidimou A. Noncontrast CT markers of intracerebral hemorrhage expansion and poor outcome: A meta-analysis. Neurology. 2020 Oct 6;95(14):632-643. doi: 10.1212/WNL.0000000000010660. Epub 2020 Aug 26. PMID 32847959
- [Background] Tseng WC, Wang YF, Wang TG, Hsiao MY. Early spot sign is associated with functional outcomes in primary intracerebral hemorrhage survivors. BMC Neurol. 2021 Mar 20;21(1):131. doi: 10.1186/s12883-021-02146-3. PMID 33743639